CLINICAL TRIAL: NCT06700512
Title: Standard PMCF Study WSA @ HZO
Brief Title: Standard Post Market Clinical Follow-up (PMCF) Study WSA @ HZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WSAUD A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D00325215
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing aid; Freiburger; Matrix Test; SSQ; IOI-HA
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Study Device followed by Own devices (Experimental): within subject design: Subjects wear the study devices for 2 weeks followed by wearing their own hearing aids for 2 weeks. Study devices are fitted as per standard-of-care.
  Interventions: Device: Hearing Aid Signia Pure C&G 7IX; Device: Own Hearing Aid

INTERVENTIONS:
Device: Hearing Aid Signia Pure C&G 7IX — Receiver in Canal (RIC) hearing aid, M Receiver
Device: Own Hearing Aid — subjects' own hearing aids, any brand, any model

SUMMARY:
The purpose of the study is to follow-up on a released low-risk device as part of standard PMCF activities

DETAILED DESCRIPTION:
This is a comparative study which is conducted monocentric at Hoerzentrum Oldenburg, Germany. The focus is to test a released hearing aid and compare this to the subject's own hearing aids with a minimum of 16 mild-to-moderate sensorineural hearing impaired adult subjects. The subjects, all of them native German speakers, have 2 appointments of 1-2 hours including a fitting procedure with real-ear measurements and some standard speech tests and undergo two 2-weeks home trials (with questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss should fall within fitting range of study hearing aid
* They should be experienced hearing aid users
* Air-Bone-Gap should be less or equal to 20 dB Hearing Loss (HL).
* Sensorineural HL, mild-to-moderate
* HL corresponding to the fitting range of the hearing aid
* Healthy (outer) ear
* Older than 18 years
* German is mother tongue
* Able to understand the instructions
* Willing to participate in laboratory tests and to wear the hearing aids at home for 2 weeks
* Informed consent

Exclusion Criteria:

* Contraindication for hearing aid treatment
* Fluctuating or rapidly progressing hearing loss
* "Central" hearing problems
* Limited mobility
* Limited dexterity (in handling the hearing aid)
* Known psychological problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Vormann, PhD, Principal Investigator — Hörzentrum Oldenburg gGmbH
Locations (1):
- Hörzentrum Oldenburg gGmbH, Oldenburg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Evaluation of Study Device Followed by Own Devices: within subject design: Subjects wear the study devices for 2 weeks followed by wearing their own hearing aids for 2 weeks. Study devices are fitted as per standard-of-care.
  Study Hearing Aid Signia Pure C&G 7IX: Receiver in Canal (RIC) hearing aid, M Receiver
  Own Hearing Aid: subjects' own hearing aids, any brand, any model
Period: Field Test 1 (2 Weeks) Study Devices
Arm/Group | Evaluation of Study Device Followed by Own Devices
Started | 20
Completed | 20
Not Completed | 0
Period: Field Test 2 (2 Weeks) Own Devices
Arm/Group | Evaluation of Study Device Followed by Own Devices
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: within subject design: compare Pure C&G 7IX to subjects' own hearing aids. Baseline measures are the same for all study participants
Arm/Group | Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 20
mild to moderate Hearing Impairment [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Oldenburg Sentence Test
Description: The Oldenburg Sentence Test (OLSA) is an audiometric test for determining the speech recognition threshold (SRT in dB). Sentences of the form name - verb - numeral - adjective - noun are used as speech material. The sequence of words is a random combination from an inventory of 50 words in total. The design of the test prevents memorization of the sentences, so the OLSA can be repeated as often as desired. For this study speech in noise recognition was measured. Noise level was 65 dB SPL played from the back, speech was presented from front. The SRT shows the signal-to-noise ratio needed for 80% speech recognition. Lower values mean better speech understanding (i.e. the speech can be quieter with respect to the noise and still be understood). There are no minimum or maximum values.
Time Frame: Estimated Time Frame 2 weeks (Test conducted at second lab session).
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Results With Study Device: within subject design: compare speech understanding with study device to speech understanding with subjects' own hearing aids or no hearing aids (unaided).
  Study devices are Signia Pure C&G 7IX Receiver-in-the-canal hearing aids with M-Receiver
- Results Unaided: Speech test without hearing aids
- Results With Own Devices: own devices are the subjects' own hearing aids, they can be any brand, any model
Arm/Group | Results With Study Device | Results Unaided | Results With Own Devices
Number analyzed (Participants) | 20 | 20 | 20
dB | -6.6 (4.5) | -1.1 (7.5) | -3.5 (5.1)
Statistical Analysis 1: Comparison: Results With Study Device vs Results Unaided; H0 (Objective 1) SRT (study HA) is either not significantly different from SRT without HAs or significantly worse than SRT without HAs. H1(Objective 1) SRT(study HA) is significantly better than SRT without HAs. A mean difference in SRT of 1 dB measured with the Oldenburg sentence test can be assumed as a typical difference in speech intelligibility to show a clinically meaningful improvement; Test type: Superiority; p < 0.001, t-test, 1 sided; paired
Statistical Analysis 2: Comparison: Results With Study Device vs Results With Own Devices; H0 (Objective 2) SRT (study HA) is significantly worse than SRT(own HAs). H1(Objective 2) There is no difference between SRT(study HA) and SRT(own HAs) or SRT (study HA) is significantly better than SRT (own HAs) SRT= Speech Reception Threshold in dB; Test type: Non-Inferiority — A mean difference in SRT of 1 dB measured with the Oldenburg sentence test (Wagener et al, 1999a-c), can be assumed as a typical difference in speech intelligibility to show a clinically meaningful improvement (Kollmeier et al, 2011). Thus if SRT with study hearing aids is 1dB or more worse than with subjects' own hearing aids and the difference is significant (p<0.05), inferiority of study hearing aid is assumed otherwise study hearing aids are considered non-inferior; p < 0.001, t-test, 1 sided — paired

2. Secondary Outcome: Freiburger Monosyllabic Speech Test
Description: To investigate speech intelligibility (SI) performance for speech at 65dB in a quiet listening situation, the Freiburger monosyllabic speech test is used which is still the gold standard for Hearing Care Professionals (HCPs) in Germany. Results are reported in Percent correct data. Minimum is 0%, maximum is 100% with higher values meaning better speech understanding.
Time Frame: Estimated Time Frame 2 weeks (Test conducted at second lab session).
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Results With Study Device | Results Unaided | Results With Own Devices
Number analyzed (Participants) | 20 | 20 | 20
Percent Correct | 75.1 (12.3) | 31.5 (20.1) | 68.6 (12.7)

3. Secondary Outcome: Match-to-Target
Description: Investigate how close the study hearing aids fitted and fine-tuned with the fitting software to NAL-NL2 Targets match the postulated targets, as measured in-situ with real-ear measurements. Absolute deviations were calculated at specific frequencies ranging from 250 Hz to 4 kHz. Unit of measure is dB SPL. Minimum Value is 0 (i.e. measured value and target value identical), no maximum value. Higher values mean greater deviation from target.
Time Frame: 1 day (Fitting procedure with real-ear measurements is done at first lab session)
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Match-to-Target Study Devices: The match-to-target was only evaluated for the study devices as an indication how well Signia hearing aids can be fitted to clinical targets (here NAL-NL2).
Arm/Group | Match-to-Target Study Devices
Number analyzed (Participants) | 20
dB
  Deviation from Target @ 250 Hz | 3.3 (4.0)
  Deviation from Target @ 500 Hz | 1.6 (1.7)
  Deviation from Target @ 1000 Hz | 1.2 (1.4)
  Deviation from Target @ 2000 Hz | 1.6 (1.9)
  Deviation from Target @ 4000 Hz | 1.5 (1.7)

4. Secondary Outcome: Speech, Spatial and Qualities of Hearing Questionnaire (SSQ)
Description: A short form of the SSQ is used (SSQ 17, German version), to investigate speech perception, sound localisation, quality of hearing perceived in real-life. Questions are answered on a scale from 0 to 10, higher scores mean better outcomes. The responses to the individual questions are grouped for the subsections (speech, spatial, quality) by calculating the means.
Time Frame: 2 weeks
Population: The aim of the SSQ questionnaire was to compare the performance/benefit of the study hearing aids to the subjects' own devices. As the unaided ratings would have been the same for both arms, they would have cancelled out by comparing the two interventions and thus it was considered as not necessary to collect the unaided responses.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- With Study Device: Results of SSQ after wearing the study devices for 2 weeks in everyday life.
- With Own Devices: Results of SSQ after wearing their own hearing aids or 2 weeks in everyday life.
Arm/Group | With Study Device | With Own Devices
Number analyzed (Participants) | 20 | 20
score on a scale
  Speech Perception | 6.2 (2.3) | 5.8 (1.9)
  Sound Localization | 6.9 (2.4) | 6.2 (1.6)
  Quality of Hearing | 7.9 (1.3) | 7.3 (1.7)

5. Secondary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA)
Description: Investigate outcomes and effectiveness of hearing aid usage in real-life. Responses are given on a scale from 1 - 5. Here, the mean of questions 2 -7 is reported. Higher values represent better outcomes. Question 1 was on wearing time, which is not considered a rating of effectiveness and was therefore excluded from the mean and will be reported separately. Fpr wearing times higher values represent longer wearing time (maximum 5 equals "more than 8 hours a day").
Time Frame: 2 weeks
Population: The IOI-HA was developed to measure outcomes in audiological rehabilitation using Hearing Aids and is not designed for the unaided condition. For this reason only the two interventional arms are included for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- With Study Device: Results of IOI-HA after wearing the study devices for 2 weeks in everyday life.
- With Own Devices: Results of IOI-HA after wearing their own hearing aids or 2 weeks in everyday life.
Arm/Group | With Study Device | With Own Devices
Number analyzed (Participants) | 20 | 20
score on a scale
  Mean effectiveness ratings | 3.6 (1.0) | 3.8 (0.7)
  Wearing Time | 5.0 (0.2) | 4.9 (0.3)

6. Secondary Outcome: Satisfaction Questionnaire
Description: Investigate satisfaction in real-life for different aspects such as sound quality, naturalness of sound, conversation with one person and overall satisfaction. Each aspect was assessed on on a 7-point likert scale, going from 1 (very dissatisfied) to 7 (very satisfied) The overall satisfaction and sound quality overall were individual questions and are not the combination of different situations/aspects. These questions were also assessed on on a 7-point likert scale, going from 1 (very dissatisfied) to 7 (very satisfied). Higher values represent better outcomes.
Time Frame: 2 weeks
Population: The satisfaction questionnaire was developed to measure satisfaction with hearing aids and not designed for the unaided condition. For this reason data was only collected for the two interventional arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- With Study Device: Results of satisfaction questionnaire after wearing the study devices for 2 weeks in everyday life.
- With Own Devices: Results of satisfaction questionnaire after wearing their own hearing aids or 2 weeks in everyday life.
Arm/Group | With Study Device | With Own Devices
Number analyzed (Participants) | 20 | 20
score on a scale
  Sound quality overall | 5.4 (1.3) | 5.5 (1.2)
  Overall Satisfaction | 5.1 (1.5) | 5.1 (1.5)
  Naturalness | 5.4 (1.4) | 5.2 (1.5)
  Conversation with one person | 5.4 (1.6) | 5.6 (1.4)
  Comfort with loud sounds | 5.0 (1.3) | 4.5 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant during the course of the study for an average time period of 4 weeks, starting with the first lab session and ending with the end of the second field test.
Groups:
- While Wearing Study Devices: Subjects wore the study devices for 2 weeks during first field test
- While Wearing Own Devices: Subjects wore their own devices for 2 weeks during second field test
Arm/Group | While Wearing Study Devices | While Wearing Own Devices
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT06700512/Prot_SAP_000.pdf